CLINICAL TRIAL: NCT02039791
Title: Phase II Study of Nimotuzumab in Combination With Neoadjuvant Chemotherapy for Cervical Cancer
Brief Title: Study of Nimotuzumab in Combination With Neoadjuvant Chemotherapy for Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-CC-072
Record Dates: First submitted 2014-01-08; First posted 2014-01-20 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nimotuzumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab plus chemoradiotherapy (Experimental)
  Interventions: Biological: Nimotuzumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Nimotuzumab — 200mg/w,weekly, 6 weeks
Drug: Carboplatin — AUC 6, d1，1 cycle/21d, 2 cycles
Drug: Paclitaxel — 175 mg/m2, d1
  1 cycle/21d, 2 cycles.

SUMMARY:
Nimotuzumab is a humanized monoclonal antibody against epidermal growth factor receptor (EGFR). Clinical trials are ongoing globally to evaluate Nimotuzumab in different indications. Nimotuzumab has been approved to treat squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal carcinoma in different countries. The clinical phaseⅡtrial is designed to assess the resection rate and pathological complete response of nimotuzumab plus carboplatin and paclitaxel in patients with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-70 years
2. Histological confirmed Cervical squamous cell carcinoma
3. FIGO Stage: IB2-IIIB
4. Tumor lesions and stages are confirmed by the internal medicine, obstetrics and gynecology inspection, including a pelvic exam and abdominal and pelvic CT,.if necessary, laparoscopy, cystoscopy and pelvic MRI examination will be taken.
5. At least one lesions can be measured
6. No previous therapy
7. ECOG performance status 0-2
8. Life expectancy of more than 6 months
9. Normal hematology:Haemoglobin≥90g/L,white blood cell(WBC)≥4×109/L Absolute neutrophil count≥1.5×109/L,platelet count≥100×109/L, normal renal function: serum creatinine<1.5mg/dl or creatinine clearance rate>60ml/min；normal liver function:TBIL≤1.5 ULN, AST and ALT≤1.5 ULN
10. Without lung or heart disease
11. Without active infection
12. Signed informed consent and submit to the organization of research

Exclusion Criteria:

1. Severe systemic or uncontrolled disease, unfit for chemotherapy
2. Neuropathy caused by any reason
3. Psychiatric disease
4. Other malignant tumor
5. Bilateral renal pelvis and ureter hydrocephalus who can't be alleviated by ureteral stent or percutaneous nephrostomy, Abnormal serum creatinine level
6. Infection and severe systemic disease
7. Received other anti EGFR monoclonal antibody treatment
8. Participation in other interventional clinical trials
9. Allergic constitution or history of drug allergy
10. Pregnant or breast-feeding or refused to take contraceptive method
11. Poor compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
resection rate | the day right after surgery
Pathological response rate | the day right after surgery

SECONDARY OUTCOMES:
objective response rate（ORR） | The first seven weeks after the end of treatment
Progression free survival progression-free survival (PFS) | Follow-up is for three consecutive years after surgery. Once every three months in the first year, and then once every six months in the second and third year.

CONTACTS AND LOCATIONS:
Overall Officials: yaping Zhu, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai first people's hospital, Shanghai, Shanghai Municipality, China